CLINICAL TRIAL: NCT05949333
Title: Reducing Neutropenia Incidence by Changing the Date of Eflapegrastim Administration in Breast Cancer Patients Who Have Experienced Neutropenia After Chemotherapy
Brief Title: Reducing Neutropenia Incidence With Pegfilgrastim Administration on Day 3 After Chemotherapy
Acronym: NEUTHREE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eunseong Medical Foundation Good GANG-AN HOSPITAL (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Changwan Jeon, Chief of Breast Center, Eunseong Medical Foundation Good GANG-AN HOSPITAL
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGAH 2022-10
Record Dates: First submitted 2023-05-30; First posted 2023-07-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — eflapegrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Day1 Group (Active Comparator): Eflapegrastim administration on day 1 (24 hours after completion of chemotherapy)
  Interventions: Drug: Eflapegrastim
- Day 3 Group (Experimental): Eflapegrastim administration on day 3 (the third day after completion of chemotherapy
  Interventions: Drug: Eflapegrastim

INTERVENTIONS:
Drug: Eflapegrastim — long-acting granulocyte-colony stimulating factor
  Other Names: Rolvedon, Eflapegrastim-xnst, HM-10460A, SPI-2012

SUMMARY:
Patients who experienced neutropenia after receiving pegfilgrastim on day 1 of the first round are randomly assigned to either the control or experimental arm. Patients in the control arm continue pegfilgrastim injection on day 1 while patients in the experimental arm will receive pegfilgrastim injection on day 3 to see if changing the pegfilgrastim administration date from day 1 to day 3 starting from the second round of chemotherapy could reduce the incidence of neutropenia

DETAILED DESCRIPTION:
The use of pegfilgrastim, which has a long-lasting effect in the human body, after myelosuppressive chemotherapy for solid tumors, including breast cancer, and blood cancers has led to a decrease in the incidence of neutropenia, including febrile neutropenia, and a reduction in medical costs by shortening hospitalization periods related to side effects of chemotherapy. During the early stages of drug development, there was controversy over the timing of pegfilgrastim administration, and attempts were made to administer it at various times, from the day of chemotherapy to the day of neutropenia began. However, based on several studies, it is now known that patients who receive pegfilgrastim on the day of chemotherapy or after 4 days of chemotherapy have a higher incidence of febrile neutropenia. Therefore, administering pegfilgrastim on day 1-3 after chemotherapy is ideal, but in reality, it is often difficult for patients to visit the hospital multiple times after chemotherapy, so many patients are discharged after receiving pegfilgrastim on day 1. The FDA and National Comprehensive Cancer Network (NCCN) guidelines also recommend administration on day 1. It is known that patients who experience neutropenia after the first round of chemotherapy are more likely to experience it again in subsequent rounds. The investigators aimed to see whether changing the pegfilgrastim administration date from day 1 to day 3 starting from the second round of chemotherapy for patients who experienced neutropenia after receiving pegfilgrastim on day 1 of the first round can reduce the incidence of neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 75 years old as of the date of study registration.
* Patients with histologically confirmed invasive adenocarcinoma.
* Patients with confirmed estrogen receptor, progesterone receptor, and Her2 receptor status.
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients with a left ventricular ejection fraction (LVEF) ≥55%.
* Patients who have agreed to participate in this trial and have provided written consent.

Exclusion Criteria:

* Patients with a history of breast cancer treatment
* Patients with a history of chemotherapy, radiation therapy, immunotherapy, or biotherapy for malignancies other than breast cancer
* Patients with infectious diseases
* Patients with serious illnesses that may affect this clinical trial: cardiovascular disease, kidney disease, liver disease, endocrine disease, tumors, or diabetes
* Other individuals deemed by the clinical trial investigators to be unable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of severe neutropenia Incidence rate of severe neutropenia | cycle 2-5 (21 days for each cycle), 105 days
  The incidence rates of Grade 4 neutropenia (ANC < 500 respectively)

SECONDARY OUTCOMES:
Duration of severe neutropenia | cycle 2-5 (21 days for each cycle), 105 days
  number of consecutive days ANC lower than 500
Incidence rate of febrile neutropenia | cycle 2-5 (21 days for each cycle), 105 days
  Severe neutropenia with fever. Fever is defined as below
  * 37.5℃ single axillary temperature
  * 38.0℃ single ear probe temperature
  * 38.3℃ single oral temperature
  * 38.0℃ oral temperature over 1 hour in the absence of an obvious cause
Incidence rate of neutropenia related death | 1 year
  Death related chemotherapy induced neutropenia sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wan Jeon, Ph.D, Principal Investigator — Surgical Oncologist
Locations (1):
- Good Gang-An Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meropol NJ, Miller LL, Korn EL, Braitman LE, MacDermott ML, Schuchter LM. Severe myelosuppression resulting from concurrent administration of granulocyte colony-stimulating factor and cytotoxic chemotherapy. J Natl Cancer Inst. 1992 Aug 5;84(15):1201-3. doi: 10.1093/jnci/84.15.1201. No abstract available. PMID 1378905
- [Background] Rowinsky EK, Grochow LB, Sartorius SE, Bowling MK, Kaufmann SH, Peereboom D, Donehower RC. Phase I and pharmacologic study of high doses of the topoisomerase I inhibitor topotecan with granulocyte colony-stimulating factor in patients with solid tumors. J Clin Oncol. 1996 Apr;14(4):1224-35. doi: 10.1200/JCO.1996.14.4.1224. PMID 8648378
- [Background] Weycker D, Bensink M, Lonshteyn A, Doroff R, Chandler D. Risk of chemotherapy-induced febrile neutropenia by day of pegfilgrastim prophylaxis in US clinical practice from 2010 to 2015. Curr Med Res Opin. 2017 Dec;33(12):2107-2113. doi: 10.1080/03007995.2017.1386858. Epub 2017 Oct 16. PMID 28958157
- [Background] Weycker D, Li X, Tzivelekis S, Atwood M, Garcia J, Li Y, Reiner M, Lyman GH. Burden of Chemotherapy-Induced Febrile Neutropenia Hospitalizations in US Clinical Practice, by Use and Patterns of Prophylaxis with Colony-Stimulating Factor. Support Care Cancer. 2017 Feb;25(2):439-447. doi: 10.1007/s00520-016-3421-x. Epub 2016 Oct 12. PMID 27734153
- [Background] Lyman GH, Allcott K, Garcia J, Stryker S, Li Y, Reiner MT, Weycker D. The effectiveness and safety of same-day versus next-day administration of long-acting granulocyte colony-stimulating factors for the prophylaxis of chemotherapy-induced neutropenia: a systematic review. Support Care Cancer. 2017 Aug;25(8):2619-2629. doi: 10.1007/s00520-017-3703-y. Epub 2017 May 8. PMID 28484882
- [Background] Kaufman PA, Paroly W, Rinaldi D. Randomized double blind phase 2 study evaluating same-day vs. next-day administration of pegfilgrastim with docetaxel, doxorubicin and cyclophosphamide (TAC) in women with early stage and advanced breast cancer. Breast Cancer Res Treat 2004;88:S59.
- [Background] Saven A, Schwartzberg L, Kaywin P, et al. Randomized, double-blind, phase 2, study evaluating same-day vs next-day administration of pegfilgrastim with R-CHOP in non-Hodgkin's lymphoma patients. J ClinOncol2006;24:7570.
- [Background] Leonard RC, Miles D, Thomas R, Nussey F; UK Breast Cancer Neutropenia Audit Group. Impact of neutropenia on delivering planned adjuvant chemotherapy: UK audit of primary breast cancer patients. Br J Cancer. 2003 Dec 1;89(11):2062-8. doi: 10.1038/sj.bjc.6601279. PMID 14647139
- [Background] Hughes WT, Armstrong D, Bodey GP, Bow EJ, Brown AE, Calandra T, Feld R, Pizzo PA, Rolston KV, Shenep JL, Young LS. 2002 guidelines for the use of antimicrobial agents in neutropenic patients with cancer. Clin Infect Dis. 2002 Mar 15;34(6):730-51. doi: 10.1086/339215. Epub 2002 Feb 13. No abstract available. PMID 11850858
- [Background] Tamura K. Clinical guidelines for the management of neutropenic patients with unexplained fever in Japan: validation by the Japan Febrile Neutropenia Study Group. Int J Antimicrob Agents. 2005 Dec;26 Suppl 2:S123-7; discussion S133-40. doi: 10.1016/j.ijantimicag.2005.08.001. Epub 2005 Oct 24. PMID 16249072